CLINICAL TRIAL: NCT00851799
Title: Cardiovascular, Anthropometric, and Skeletal Effects of Antiretroviral Therapy (ART) Initiation With Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) Plus Atazanavir/Ritonavir (ATV/r), Darunavir/Ritonavir (DRV/r), or Raltegravir (RAL): Metabolic Substudy of A5257
Brief Title: Impact of Antiretroviral Therapy on Metabolic, Skeletal, and Cardiovascular Parameters
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5260s; 1U01AI068636 (NIH); ACTG A5257 metabolic substudy
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infection
Keywords: ART; Antiretroviral therapy; Treatment naive; Highly active antiretroviral therapy (HAART)
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ritonavir; Atazanavir Sulfate; Raltegravir Potassium; Darunavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples will be collected and stored

GROUPS / COHORTS (3):
- Cohort A: ATV/RTV + FTC/TDF
  Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF), ritonavir (RTV), and atazanavir (ATV) to be taken orally, once daily.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Ritonavir; Drug: Atazanavir
- Cohort B: RAL + FTC/TDF
  FTC/TDF orally, once daily, and raltegravir (RAL) orally, twice daily.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Ritonavir; Drug: Raltegravir
- Cohort C: DRV/RTV + FTC/TDF
  FTC/TDF, darunavir (DRV), and RTV, orally, once daily.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Ritonavir; Drug: Darunavir

INTERVENTIONS:
Drug: Emtricitabine/tenofovir disoproxil fumarate — 200 mg emtricitabine/300 mg tenofovir disoproxil fumarate taken orally daily. A combination drug of two nucleoside reverse transcriptase inhibitors (NRTIs).
  Other Name: TDF/FTC
Drug: Ritonavir — 100 mg taken orally once daily. A protease inhibitor (PI).
  Other Name: RTV
Drug: Atazanavir — 300 mg taken orally once daily. A protease inhibitor (PI).
  Other Name: ATV
  Groups: Cohort A
Drug: Raltegravir — 400 mg taken orally twice daily. An integrase inhibitor (INI).
  Other Name: RAL
  Groups: Cohort B
Drug: Darunavir — 100 mg taken orally once daily. A protease inhibitor (PI).
  Other Name: RTV
  Groups: Cohort C

SUMMARY:
The U.S. Department of Health and Human Services (HHS) guidelines recommend that HIV-infected people who have never received anti-HIV therapy be treated with a triple drug regimen (commonly called combination antiretroviral therapy, cART). Since the introduction of cART, morbidity and mortality among HIV-infected patients has been dramatically reduced. However, metabolic, skeletal, and cardiovascular diseases have been increasingly reported among HIV-infected patients and may be attributable, in part, to the direct effects of cART. Much of our understanding of the development of these diseases, risk factors, and consequences of these disorders has been derived from clinical studies of HIV-infected persons receiving older antiretroviral agents.

A5260s was designed to examine the contributions of HIV-disease related factors and impact of newer antiretroviral drugs on the development of metabolic (such as blood vessels, blood sugar, cholesterol), skeletal, and cardiovascular diseases in people who have never received anti-HIV therapy. A5260s is a prospective substudy of a phase III randomized clinical trial A5257 (see ClinicalTrials.gov identifier: NCT00811954). A5257 was designed to look at different combinations of anti-HIV drugs that do not contain the medication efavirenz (EFV) and how well these drug combinations work to decrease the amount of HIV in the blood and to allow immune system recovery in people who have never received anti-HIV therapy. A5257 also examined drug tolerability and safety for the various drug combinations.

DETAILED DESCRIPTION:
A5260s is the optional, metabolic substudy of a phase III, prospective, randomized clinical trial (A5257). For complete details about the parent study A5257, please see ClinicalTrials.gov identifier NCT00811954.

Some participants in study A5257 were asked to participate in substudy A5260s. Not all participants were asked since A5260s only took place at a subset of A5257 sites. Participants who agreed to participate in substudy A5260s were enrolled at the same time as their enrollment in A5257. No interventions were given as part of A5260s, but all A5260s participants underwent blood draws, self-administered questionnaire responses (related to physical activity and body image), ultrasound scans to measure the thickness of the carotid artery in the neck and brachial artery flow mediated dilation in the arm, and computerized topography (CT) and dual-energy x-ray absorptiometry (DEXA) scans to measure bone mineral density and body fat.

The duration of A5260s study was between 2 and 3 years (96 and 144 weeks), depending on when the participant enrolled. The study was designed to enroll a total of 330 participants with at least 110 per a group; each group represented a different randomized drug combination as defined and assigned by the main study A5257.

Cohort A: Atazanavir (ATV) + Ritonavir (RTV) + Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF)

Cohort B: Raltegravir (RAL) + FTC/TDF

Cohort C: Darunavir (DRV) + RTV + FTC/TDF

All participants were asked to return for A5260s clinic visits at weeks 4, 24, 48 96 and 144 and participated in all clinical evaluations. No clinical evaluation was restricted to a subset of A5260s participants. If a participant chose to discontinue participation in the substudy, the participant was able to continue in study A5257. However, a participant discontinuing participation from A5257 was also removed from A5260s. Additionally, a participant's decision to discontinue or switch study drugs in the main study did not impact participation and follow-up clinic visits in A5260s.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in A5257 and intent to enroll in A5001 (ALLRT)
* Signed informed consent
* For A5257 inclusion criteria, please see ClinicalTrials.gov identifier NCT00811954

Exclusion Criteria:

* Diabetes mellitus, (fasting plasma glucose ≥ 126 mg/dL on two occasions or on hypoglycemic medications).
* Known cardiovascular disease (history of myocardial infarction [MI], coronary artery bypass graft surgery, percutaneous coronary intervention, stroke, transient ischemic attack, or peripheral arterial disease with ankle-brachial index of less than 0.9 or claudication)
* Uncontrolled hypothyroidism or hyperthyroidism which in the opinion of the site investigator would affect substudy participation
* Current use of statins, fish oil (greater than 2 grams per day), fibric acid derivatives, or niacin (more than 1000 mg per day) (NOTE: Current use of fish oil and niacin is defined as receiving treatment in the 8 weeks prior to study entry)
* Intention to start pharmacological or surgical intervention for weight loss
* Use of any ART in the 30 days before study entry
* For A5257 exclusion criteria, please see ClinicalTrials.gov identifier NCT00811954

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Antiretroviral naïve, HIV-infected men and women with HIV-1 RNA level >1000 copies/ml initiating treatment for HIV-1 infection.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Brown, MD, PhD, Study Chair — Johns Hopkins University; James Stein, MD, Study Chair — University of Wisconsin, Madison; Grace McComsey, MD, FIDSA, Study Chair — University Hospitals Cleveland Medical Center; Judith Currier, MD, MSc, Study Chair — UCLA AIDS Prevention & Treatment CTU
Locations (26):
- United States (26):
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor - UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - The Ponce de Leon Center, Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush University Medical Center (2702), Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Washington University CRS (2101), St Louis, Missouri
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - AIDS Care CRS, Rochester, New York
  - University of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS (1601), Durham, North Carolina
  - University of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - Metro Health CRS, Cleveland, Ohio
  - The Ohio State University AIDS CRS (2301), Colombus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington

REFERENCES:
- [Background] Lennox JL, Landovitz RJ, Ribaudo HJ, Ofotokun I, Na LH, Godfrey C, Kuritzkes DR, Sagar M, Brown TT, Cohn SE, McComsey GA, Aweeka F, Fichtenbaum CJ, Presti RM, Koletar SL, Haas DW, Patterson KB, Benson CA, Baugh BP, Leavitt RY, Rooney JF, Seekins D, Currier JS; ACTG A5257 Team. Efficacy and tolerability of 3 nonnucleoside reverse transcriptase inhibitor-sparing antiretroviral regimens for treatment-naive volunteers infected with HIV-1: a randomized, controlled equivalence trial. Ann Intern Med. 2014 Oct 7;161(7):461-71. doi: 10.7326/M14-1084. PMID 25285539
- [Background] Ofotokun I, Na LH, Landovitz RJ, Ribaudo HJ, McComsey GA, Godfrey C, Aweeka F, Cohn SE, Sagar M, Kuritzkes DR, Brown TT, Patterson KB, Para MF, Leavitt RY, Villasis-Keever A, Baugh BP, Lennox JL, Currier JS; AIDS Clinical Trials Group (ACTG) A5257 Team. Comparison of the metabolic effects of ritonavir-boosted darunavir or atazanavir versus raltegravir, and the impact of ritonavir plasma exposure: ACTG 5257. Clin Infect Dis. 2015 Jun 15;60(12):1842-51. doi: 10.1093/cid/civ193. Epub 2015 Mar 12. PMID 25767256
- [Background] Vardhanabhuti S, Ribaudo HJ, Landovitz RJ, Ofotokun I, Lennox JL, Currier JS, Olson LM, Haas DW. Screening for UGT1A1 Genotype in Study A5257 Would Have Markedly Reduced Premature Discontinuation of Atazanavir for Hyperbilirubinemia. Open Forum Infect Dis. 2015 Jul 1;2(3):ofv085. doi: 10.1093/ofid/ofv085. eCollection 2015 Sep. PMID 26180834
- [Result] Stein JH, Ribaudo HJ, Hodis HN, Brown TT, Tran TT, Yan M, Brodell EL, Kelesidis T, McComsey GA, Dube MP, Murphy RL, Currier JS. A prospective, randomized clinical trial of antiretroviral therapies on carotid wall thickness. AIDS. 2015 Sep 10;29(14):1775-83. doi: 10.1097/QAD.0000000000000762. PMID 26372383
- [Result] Kelesidis T, Tran TT, Stein JH, Brown TT, Moser C, Ribaudo HJ, Dube MP, Murphy R, Yang OO, Currier JS, McComsey GA. Changes in Inflammation and Immune Activation With Atazanavir-, Raltegravir-, Darunavir-Based Initial Antiviral Therapy: ACTG 5260s. Clin Infect Dis. 2015 Aug 15;61(4):651-60. doi: 10.1093/cid/civ327. Epub 2015 Apr 22. PMID 25904376
- [Result] Brown TT, Moser C, Currier JS, Ribaudo HJ, Rothenberg J, Kelesidis T, Yang O, Dube MP, Murphy RL, Stein JH, McComsey GA. Changes in Bone Mineral Density After Initiation of Antiretroviral Treatment With Tenofovir Disoproxil Fumarate/Emtricitabine Plus Atazanavir/Ritonavir, Darunavir/Ritonavir, or Raltegravir. J Infect Dis. 2015 Oct 15;212(8):1241-9. doi: 10.1093/infdis/jiv194. Epub 2015 May 5. PMID 25948863
- [Result] Stein JH, Brown TT, Ribaudo HJ, Chen Y, Yan M, Lauer-Brodell E, McComsey GA, Dube MP, Murphy RL, Hodis HN, Currier JS. Ultrasonographic measures of cardiovascular disease risk in antiretroviral treatment-naive individuals with HIV infection. AIDS. 2013 Mar 27;27(6):929-937. doi: 10.1097/QAD.0b013e32835ce27e. PMID 23196938
- [Result] Brown TT, Chen Y, Currier JS, Ribaudo HJ, Rothenberg J, Dube MP, Murphy R, Stein JH, McComsey GA. Body composition, soluble markers of inflammation, and bone mineral density in antiretroviral therapy-naive HIV-1-infected individuals. J Acquir Immune Defic Syndr. 2013 Jul 1;63(3):323-30. doi: 10.1097/QAI.0b013e318295eb1d. PMID 23591634
- [Derived] Hughey CM, Vuong BW, Ribaudo HB, Mitchell CCK, Korcarz CE, Hodis HN, Currier JS, Stein JH. Grayscale Ultrasound Texture Features of Carotid and Brachial Arteries in People With HIV Infection Before and After Antiretroviral Therapy. J Am Heart Assoc. 2022 Mar;11(5):e024142. doi: 10.1161/JAHA.121.024142. Epub 2022 Feb 18. PMID 35179037
- [Derived] Debroy P, Lake JE, Moser C, Olefsky M, Erlandson KM, Scherzinger A, Stein JH, Currier JS, Brown TT, McComsey GA. Antiretroviral Therapy Initiation Is Associated With Decreased Visceral and Subcutaneous Adipose Tissue Density in People Living With Human Immunodeficiency Virus. Clin Infect Dis. 2021 Mar 15;72(6):979-986. doi: 10.1093/cid/ciaa196. PMID 32107532
- [Derived] McComsey GA, Moser C, Currier J, Ribaudo HJ, Paczuski P, Dube MP, Kelesidis T, Rothenberg J, Stein JH, Brown TT. Body Composition Changes After Initiation of Raltegravir or Protease Inhibitors: ACTG A5260s. Clin Infect Dis. 2016 Apr 1;62(7):853-62. doi: 10.1093/cid/ciw017. Epub 2016 Jan 20. PMID 26797215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consented and enrolled at AIDS clinical trials units in the United States. Enrollment occurred between June 1, 2009 (date first participant was enrolled) and April 13, 2011 (date last subject was enrolled).
Pre-assignment Details: 334 consented and enrolled; 6 participants who initially enrolled were subsequently found ineligible and excluded from all analyses. Results reported for 328 eligible participants.
Groups:
- Cohort A: ATV/RTV + FTC/TDF: ATV/RTV + FTC/TDF
  Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF), ritonavir (RTV), and atazanavir (ATV) to be taken orally, once daily.
  Emtricitabine/tenofovir disoproxil fumarate: A combination drug of two nucleoside reverse transcriptase inhibitors (NRTIs) Ritonavir: A protease inhibitor (PI) Atazanavir: A protease inhibitor (PI)
- Cohort B: RAL + FTC/TDF: RAL + FTC/TDF
  FTC/TDF orally, once daily, and raltegravir (RAL) orally, twice daily.
  Emtricitabine/tenofovir disoproxil fumarate: A combination drug of two nucleoside reverse transcriptase inhibitors (NRTIs) Raltegravir: An integrase inhibitor (INI)
- Cohort C: DRV/RTV + FTC/TDF: DRV/RTV + FTC/TDF
  FTC/TDF, darunavir (DRV), and RTV, orally, once daily.
  Emtricitabine/tenofovir disoproxil fumarate: A combination drug of two nucleoside reverse transcriptase inhibitors (NRTIs) Darunavir: A protease inhibitor (PI) Ritonavir: A protease inhibitor (PI)
Period: Overall Study
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Started | 109 | 106 | 113
Completed | 93 | 93 | 89
Not Completed | 16 | 13 | 24
Not completed — Death | 1 | 0 | 1
Not completed — Lost to Follow-up | 5 | 3 | 10
Not completed — Not able to get to clinic | 8 | 5 | 9
Not completed — Not willing to adhere to requirements | 1 | 2 | 2
Not completed — Withdrew consent prior study completion | 1 | 2 | 1
Not completed — Severe Debilitation | 0 | 1 | 0
Not completed — Completed protocol due to pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All eligible participants were included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF | Total
Number analyzed (Participants) | 109 | 106 | 113 | 328
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 107 | 105 | 113 | 325
  >=65 years | 2 | 1 | 0 | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [31 to 45] | 36 [27 to 44] | 35 [27 to 46] | 36 [28 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 12 | 34
  Male | 99 | 94 | 101 | 294
Race/Ethnicity, Customized [Number; unit: participants] — Race/Ethnicity was collected prior to study entry.
  participants
    White Non-Hispanic | 53 | 43 | 48 | 144
    Black Non-Hispanic | 34 | 34 | 37 | 105
    Hispanic (Regardless of Race) | 20 | 20 | 25 | 65
    Asian, Pacific Islander | 2 | 5 | 1 | 8
    American Indian, Alaskan Native | 0 | 2 | 1 | 3
    More than one race | 0 | 1 | 1 | 2
    Unknown/missing | 0 | 1 | 0 | 1
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] — HIV-1 RNA was calculated as the geometric mean of the two most recent HIV-1 RNA (log 10 copies/mL) obtained on or before study entry. In the event that these two values differed by more than 1 log10 copy/mL, the outlying value (based on review of all HIV-1 RNA levels available prior to study entry by the study virologist) was excluded with the baseline level determined by the remaining sample. Note that screening HIV-1 RNA values were not used in the calculation of baseline HIV-1 RNA levels.
  log10 copies/mL | 4.6 [4.0 to 5.1] | 4.5 [4.1 to 5.1] | 4.5 [4.0 to 4.9] | 4.5 [4.0 to 5.1]
CD4+ T-cell count [Median (Inter-Quartile Range); unit: cells/mm^3]] — CD4+ T-cell counts were calculated as the mean of the two most recent values available on or before study entry.
  cells/mm^3] | 350 [211 to 461] | 343 [185 to 445] | 355 [207 to 461] | 349 [203 to 455]

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Change in Right Common Carotid Artery Intima-media Thickness (CIMT)
Description: Right common carotid artery intima-media thickness was measured by ultrasound scan at study entry and weeks 48, 96 and 144.
  The annual rate of change in right common carotid artery intima-media thickness (CIMT) was estimated over 144 weeks from study entry using mixed effects linear regression model that adjusted for screening HIV-1 RNA level and Framingham risk score stratification factors.
Time Frame: Study entry, week 144
Population: Intention to treat; all eligible participants were included in the analysis. Participants were analyzed per original assigned randomized treatment and stratification in ACTG A5257.
Measure: Mean (95% Confidence Interval); unit: micron/year
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 106 | 113
micron/year | 8.2 [5.6 to 10.8] | 10.7 [9.2 to 12.2] | 12.9 [10.3 to 15.5]
Statistical Analysis 1: Comparison: Cohort A: ATV/RTV + FTC/TDF vs Cohort C: DRV/RTV + FTC/TDF; The primary hypothesis was that rate of change of CIMT would be faster over 144 weeks in participants initiating a RTV-boosted protease inhibitor-containing regimen (the pooled ATV/RTV and DRV/RTV groups) compared with a RAL-containing regimen. However, In the event of a significant difference between ATV/RTV and DRV/RTV groups, the study was designed to make all pairwise treatment group comparisons; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — Inference was assessed against a type I error of 2.5% to account for multiple comparisons; Difference in annual rate of change = -4.7, 97.5% CI 2-sided [-8.9 to -0.4] — The difference in the rate of CIMT change (Cohort A: ATV/RTV + FTC/TDF - Cohort C: DRV/RTV + FTC/TDF) was estimated by mixed effects linear regression model that adjusted for screening HIV-1 RNA level and Framingham risk score stratification factors
Statistical Analysis 2: Comparison: Cohort A: ATV/RTV + FTC/TDF vs Cohort B: RAL + FTC/TDF; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.15, Mixed Models Analysis — Inference was assessed against a type I error of 2.5% to account for multiple comparisons; Difference in annual rate of change = -2.8, 97.5% CI 2-sided [-7.0 to 1.5] — The difference in the rate of CIMT change (Cohort A: ATV/RTV + FTC/TDF - Cohort B: RAL + FTC/TDF) was estimated by mixed effects linear regression model that adjusted for screening HIV-1 RNA level and Framingham risk score stratification factors
Statistical Analysis 3: Comparison: Cohort B: RAL + FTC/TDF vs Cohort C: DRV/RTV + FTC/TDF; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.31, Mixed Models Analysis — Inference was assessed against a type I error of 2.5% to account for multiple comparisons; Difference in annual rate of change = 1.9, 97.5% CI 2-sided [-2.4 to 6.2] — The difference in the rate of CIMT change (Cohort C: DRV/RTV + FTC/TDF - Cohort B: RAL + FTC/TDF) was estimated by mixed effects linear regression model that adjusted for screening HIV-1 RNA level and Framingham risk score stratification factors

2. Primary Outcome: Change in Brachial Artery (BA) Flow Mediated Dilation (FMD) From Study Entry to Week 24
Description: Brachial artery flow mediated dilation was measured by brachial artery reactivity tests. All results reflect measures captured from participants who reported fasting and not smoking for at least 8 hours prior to FMD assessments.
  The change from study entry to week 24 in brachial artery FMD (%) was defined as the maximum FMD (%) calculated from resting heart rate (RH) 60 seconds and RH 90 seconds, relative to resting brachial artery diameter.
Time Frame: Study entry, week 24
Population: Intention to treat; all eligible participants with available data were included. Participants were analyzed per original assigned randomized treatment and stratification in ACTG A5257.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 103 | 102 | 107
percent | -0.05 [-1.51 to 1.60] | -0.27 [-1.61 to 1.55] | 0.15 [-1.39 to 1.56]
Statistical Analysis 1: Comparison: Cohort A: ATV/RTV + FTC/TDF vs Cohort C: DRV/RTV + FTC/TDF; The study was designed to compare change from study entry to week 24 in brachial artery (BA) flow mediated dilation (FMD) between a RTV-boosted protease inhibitor-containing regimen (the pooled ATV/RTV and DRV/RTV groups) and a RAL-containing regimen. However, in the event of a significant difference between ATV/RTV and DRV/RTV groups, the study was designed to make all pairwise treatment group comparisons; Test type: Superiority or Other; p = 0.53, Regression, Linear — Inference was assessed against a type I error of 2.5% to account for multiple comparisons; Difference in Change = 0.24, 97.5% CI 2-sided [-0.63 to 1.11] — The difference in change in relative FMD (Cohort A: ATV/RTV+FTC/TDF - Cohort C: DRV/RTV+FTC/TDF); estimated by linear regression that adjusted for study entry BA diameter and screening HIV-1 RNA level and Framingham risk score stratification factors
Statistical Analysis 2: Comparison: Cohort A: ATV/RTV + FTC/TDF vs Cohort B: RAL + FTC/TDF vs Cohort C: DRV/RTV + FTC/TDF; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.53, Regression, Linear — Inference was assessed against a type I error of 2.5% to account for multiple comparisons; Difference in Change (%) = -0.21, 97.5% CI 2-sided [-0.98 to 0.55] — The difference in change in relative FMD (Cohort B - Cohort A and C); estimated by linear regression that adjusted for study entry BA diameter and screening HIV-1 RNA level and Framingham risk score stratification factors

3. Secondary Outcome: Change in Brachial Artery Flow Mediated Dilation (FMD) From Study Entry to Weeks 4 and 48
Description: Brachial artery flow mediated dilation was measured by brachial artery reactivity tests. All results reflect measures captured from participants who reported fasting and not smoking for at least 8 hours prior to FMD assessments.
  The change from study entry to weeks 4 and 48 in brachial artery FMD (%) was defined as the maximum FMD (%) calculated from resting heart rate (RH) 60 seconds and RH 90 seconds, relative to resting brachial artery diameter.
Time Frame: Study entry, weeks 4 and 48
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 103 | 102 | 107
percent
  Change from study entry to week 4 | -0.04 [-0.54 to 0.46] | 0.22 [-0.36 to 0.81] | -0.15 [-0.65 to 0.34]
  Change from study entry to week 48 | -0.04 [-0.60 to 0.52] | -0.08 [-0.73 to 0.58] | -0.11 [-0.71 to 0.49]

4. Secondary Outcome: Change in Absolute Flow Mediated Dilation (FMD) From Study Entry to Weeks 4, 24 and 48
Description: The change in absolute FMD was defined as the maximum absolute FMD from the RH 60 and 90 second measurements, from study entry to weeks 4, 24, and 48 (unit of measure millimeters). All results reflect measures captured from participants who reported fasting and not smoking for at least 8 hours prior to FMD assessments.
Time Frame: Study entry, weeks 4, 24 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 103 | 102 | 107
mm
  Change from study entry to week 4 | 0.002 (0.100) | 0.012 (0.105) | -0.005 (0.102)
  Change from study entry to week 24 | -0.002 (0.103) | -0.004 (0.101) | 0.008 (0.116)
  Change from study entry to week 48 | 0.002 (0.111) | 0.005 (0.120) | -0.001 (0.119)

5. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) of the Hip From Study Entry to Week 96
Description: Bone mineral density (BMD) of the hip was evaluated by dual-energy x-ray absorptiometry (DXA) scans at study entry and study week 96. The percent change was calculated as ((week 96 value - study entry value) / study entry value)) x 100.
Time Frame: Study entry, week 96
Population: Intention to treat; all eligible participants with available data were included in the analysis. Participants were analyzed per original assigned randomized treatment and stratification in ACTG A5257
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 98 | 94 | 96
percent | -3.7 [-5.7 to -1.4] | -2.2 [-4.5 to 0.4] | -3.3 [-5.2 to -0.9]

6. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) of the Lumber Spine From Study Entry to Week 96
Description: Bone mineral density (BMD) of the lumber spine was evaluated by dual-energy x-ray absorptiometry (DXA) scans at study entry and study week 96. The percent change was calculated as ((week 96 value - study entry value) / study entry value)) x 100.
Time Frame: Study entry, week 96
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 99 | 94 | 96
percent | -4.0 [-6.5 to -0.3] | -1.6 [-3.6 to 0.9] | -3.1 [-5.2 to -0.8]

7. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) of the Total Body From Study Entry to Week 96
Description: Bone mineral density (BMD) of the total body was evaluated by dual-energy x-ray absorptiometry (DXA) scans at study entry and study week 96. The percent change was calculated as ((week 96 value - study entry value) / study entry value)) x 100.
Time Frame: Study entry, week 96
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 98 | 94 | 97
percent | -1.9 [-3.7 to -1.0] | -0.9 [-2.7 to 0.6] | -1.0 [-2.3 to 0.5]

8. Secondary Outcome: Percent Change in Total Limb Fat From Study Entry to Week 96
Description: Total limb fat was evaluated by dual-energy x-ray absorptiometry (DXA) scans at study entry and week 96. The percent change was calculated as ((week 96 value - study entry value) / study entry value)) x 100.
Time Frame: Study entry, week 96
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 98 | 94 | 97
percent | 9.8 [-3.7 to 21.3] | 6.3 [-7.5 to 27.7] | 7.9 [-5.8 to 22.9]

9. Secondary Outcome: Percent Change in Trunk Fat From Study Entry to Week 96
Description: Trunk fat was evaluated by dual-energy x-ray absorptiometry (DXA) scans at study entry and week 96. The percent change was calculated as ((week 96 value - study entry value) / study entry value)) x 100.
Time Frame: Study entry, week 96
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 98 | 94 | 97
percent | 10.8 [-3.4 to 27.7] | 13.5 [-5.3 to 38.3] | 9.7 [-3.7 to 33.6]

10. Secondary Outcome: Percent Change in Lean Mass From Study Entry to Week 96
Description: Lean mass was evaluated by dual-energy x-ray absorptiometry (DXA) scans at study entry and week 96. The percent change was calculated as ((week 96 value - study entry value) / study entry value)) x 100.
Time Frame: Study entry, week 96
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 98 | 94 | 97
percent | 1.8 [-1.2 to 4.7] | 1.7 [-1.8 to 5.0] | 0.1 [-2.1 to 2.8]

11. Secondary Outcome: Percent Change in Visceral Abdominal Fat (VAT) From Study Entry to Week 96
Description: Visceral abdominal fat (VAT) was evaluated by single slice abdominal computerized tomography scans at study entry and week 96. The percent change was calculated as as ((week 96 value - study entry value) / study entry value)) x 100.
Time Frame: Study entry, week 96
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 97 | 95 | 94
percent | 10.7 [-12.0 to 50.2] | 16.2 [-7.9 to 43.3] | 9.5 [-8.7 to 37.8]

12. Secondary Outcome: Percent Change in Subcutaneous Abdominal Fat (SAT) From Study Entry to Week 96
Description: Subcutaneous abdominal fat (SAT) was evaluated by single slice abdominal computerized tomography scans at study entry and week 96. The percent change was calculated as ((week 96 value - study entry value) / study entry value)) x 100.
Time Frame: Study entry, week 96
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 97 | 95 | 94
percent | 10.3 [-5.9 to 26.5] | 11.8 [-6.5 to 36.1] | 11.4 [-7.9 to 33.4]

13. Secondary Outcome: CD4+ T-cell Count at Study Entry and Weeks 24, 48, 96 and 144
Description: The absolute levels of CD4+ T-cell counts (cells/mm^3) measured at study entry and weeks 24, 48, 96 and 144.
Time Frame: Study entry, weeks 24, 48, 96 and 144
Population: Intention to treat; all eligible participants with available data were included. Missing data were assumed missing completely at random. Participants were analyzed per original assigned randomized treatment in ACTG A5257.
Measure: Median (Inter-Quartile Range); unit: cell/mm^3
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 106 | 113
cell/mm^3
  Study Entry | 350 [211 to 461] | 343 [185 to 445] | 355 [207 to 461]
  Week 24 | 509 [356 to 653] | 445 [348 to 610] | 464 [299 to 592]
  Week 48 | 573 [414 to 716] | 496 [367 to 689] | 528 [355 to 627]
  Week 96 | 634 [452 to 768] | 569 [416 to 717] | 567 [417 to 749]
  Week 144 | 658 [478 to 834] | 613 [437 to 801] | 560 [431 to 756]

14. Secondary Outcome: Change in CD4+ T-cell Count From Study Entry to Weeks 24, 48, 96 and 144
Description: Change was calculated as (CD4+ T-cell count at week 24, 48, 96, or 144) - (CD4+ T-cell count at study entry).
Time Frame: Study entry to weeks 24, 48, 96, and 144
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: cell/mm^3
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 107 | 99 | 108
cell/mm^3
  Change from study entry to week 24 | 161 [91 to 252] | 133 [63 to 216] | 118 [33 to 203]
  Change from study entry to week 48 | 209 [138 to 319] | 191 [89 to 311] | 194 [76 to 276]
  Change from study entry to week 96 | 280 [180 to 390] | 247 [107 to 343] | 248 [124 to 341]
  Change from study entry to week 144 | 305 [209 to 426] | 279 [142 to 400] | 227 [115 to 391]

15. Secondary Outcome: Change in Fasting Total Cholesterol (TC) From Study Entry to Weeks 4, 24, 48 and 96
Description: Total cholesterol (TC, unit of measure mg/dL) was measured at study entry and weeks 4, 24, 48 and 96 from participants who reported fasting for at least 8 hours prior to assessment; all results were centrally laboratory tested in batch. Change in TC was calculated as (week 4, 24, 48 or 96 result) - (study entry result).
Time Frame: Study entry, weeks 4, 24, 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 105 | 112
mg/dL
  Change from study entry to week 4 | 4 [-11 to 19] | -7 [-25 to 9] | 3 [-13 to 21]
  Change from study entry to week 24 | 9 [-8 to 24] | -4 [-23 to 14] | 7 [-6 to 33]
  Change from study entry to week 48 | 8 [-8 to 26] | -1 [-24 to 24] | 12 [-7 to 31]
  Change from study entry to week 96 | 12 [-6 to 32] | 1 [-16 to 23] | 14 [-8 to 38]

16. Secondary Outcome: Change in Fasting Triglyceride (TG) From Study Entry to Weeks 4, 24, 48 and 96
Description: Triglyceride (TG, unit of measure mg/dL) was measured at study entry and weeks 4, 24, 48 and 96 from participants who reported fasting for at least 8 hours prior to assessment; all results were centrally laboratory tested in batch. Change in TG was calculated as (week 4, 24, 48 or 96 result) - (study entry result).
Time Frame: Study entry, weeks 4, 24, 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 105 | 112
mg/dL
  Change from study entry to week 4 | 14 [-19 to 50] | -12 [-41 to 11] | 15 [-7 to 43]
  Change from study entry to week 24 | 6 [-20 to 39] | -16 [-48 to 4] | 2 [-19 to 46]
  Change from study entry to week 48 | 9 [-22 to 50] | -13 [-40 to 13] | 8 [-18 to 41]
  Change from study entry to week 96 | 10 [-29 to 45] | -7 [-28 to 19] | 0 [-27 to 28]

17. Secondary Outcome: Change in Fasting High-density Lipoprotein Cholesterol (HDL-C) From Study Entry to Weeks 4, 24, 48 and 96
Description: HDL cholesterol (unit of measure mg/dL) was measured at study entry and weeks 4, 24, 48 and 96 from participants who reported fasting for at least 8 hours prior to assessment; all results were centrally laboratory tested in batch. Change in HDL-C was calculated as (week 4, 24, 48 or 96 result) - (study entry result).
Time Frame: Study entry, weeks 4, 24, 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 105 | 112
mg/dL
  Change from study entry to week 4 | -1 [-6 to 6] | -2 [-6 to 4] | -3 [-7 to 2]
  Change from study entry to week 24 | 3 [-3 to 10] | 3 [-4 to 7] | 0 [-5 to 9]
  Change from study entry to week 48 | 2 [-5 to 10] | 2 [-3 to 10] | 1 [-3 to 6]
  Change from study entry to week 96 | 4 [-3 to 10] | 4 [-2 to 10] | 4 [-3 to 9]

18. Secondary Outcome: Change in Fasting Calculated Low-density Lipoprotein Cholesterol (LDL-C) From Study Entry to Weeks 4, 24, 48 and 96
Description: Calculated LDL-C (unit of measure mg/dL) was measured at study entry and weeks 4, 24, 48 and 96 from participants who reported fasting for at least 8 hours prior to assessment; all results were centrally laboratory tested in batch. Change in calculated LDL-C was calculated as (week 4, 24, 48 or 96 result) - (study entry result).
Time Frame: Study entry, weeks 4, 24, 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 108 | 104 | 110
mg/dL
  Change from study entry to week 4 | 0 [-12 to 11] | -3 [-17 to 10] | 1 [-6 to 17]
  Change from study entry to week 24 | 2 [-15 to 16] | -2 [-16 to 14] | 3 [-8 to 24]
  Change from study entry to week 48 | 1 [-12 to 17] | -1 [-16 to 21] | 5 [-8 to 19]
  Change from study entry to week 96 | 2 [-11 to 20] | -1 [-15 to 18] | 6 [-8 to 31]

19. Secondary Outcome: Change in Fasting Glucose Level From Study Entry to Weeks 4, 24, 48 and 96
Description: Glucose (unit of measure mg/dL) was measured at study entry and weeks 4, 24, 48 and 96; all results reflect measures captured from participants who reported fasting for at least 8 hours prior to assessment. Change was calculated as (fasting result during at week 4, 24, 48 or 96) - (fasting result at study entry).
Time Frame: Study entry, weeks 4, 24, 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 105 | 112
mg/dL
  Change from study entry to week 4 | 3 [-2 to 8] | 3 [-2 to 8] | 2 [-3 to 7]
  Change from study entry to week 24 | 4 [-1 to 8] | 4 [0 to 10] | 4 [-3 to 8]
  Change from study entry to week 48 | 4 [-2 to 14] | 4 [-2 to 10] | 2 [-5 to 7]
  Change from study entry to week 96 | 3 [-2 to 10] | 6 [2 to 13] | 2 [-2 to 8]

20. Secondary Outcome: Change in Fasting Insulin Level From Study Entry to Weeks 4, 24, 48 and 96
Description: Insulin (unit of measure uIU/dL) was measured at study entry and weeks 4, 24, 48 and 96; all results reflect measures captured from participants who reported fasting for at least 8 hours prior to assessment. Change was calculated as (fasting result during at week 4, 24, 48 or 96) - (fasting result at study entry).
Time Frame: Study entry, weeks 4, 24, 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: uIU/dL
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 105 | 112
uIU/dL
  Change from study entry to week 4 | 4.0 [1.0 to 8.0] | 3.0 [0.0 to 6.0] | 3.0 [0.0 to 5.0]
  Change from study entry to week 24 | 4.0 [1.0 to 8.0] | 3.0 [1.0 to 5.0] | 2.0 [0.0 to 6.0]
  Change from study entry to week 48 | 4.0 [0.0 to 9.0] | 3.0 [0.0 to 7.0] | 3.0 [0.0 to 5.0]
  Change from study entry to week 96 | 3.5 [0.0 to 8.0] | 3.0 [0.0 to 6.0] | 2.0 [0.0 to 6.0]

21. Secondary Outcome: Fold Change in D-dimer From Study Entry to Weeks 48 and 96
Description: D-dimer was measured at study entry and weeks 48 and 96 (unit of measure ug/ml). Fold change from study entry to week 48 or week 96 was calculated as (week 48 value or week 96 value) / (study entry value). Results identified above or below the limit of quantification were imputed at the quantification limit of the respective assay.
Time Frame: Study entry, weeks 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold change
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 108 | 105 | 110
Fold change
  Fold change from study entry to week 48 | 0.57 [0.31 to 1.00] | 0.73 [0.40 to 1.43] | 0.65 [0.35 to 1.00]
  Fold change from study entry to week 96 | 0.52 [0.26 to 1.00] | 0.72 [0.44 to 1.15] | 0.65 [0.29 to 1.53]

22. Secondary Outcome: Fold Change in High Sensitivity C-reactive Protein (hsCRP) From Study Entry to Weeks 48 and 96
Description: hsCRP was measured at study entry and weeks 48 and 96 (unit of measure ug/ml). Fold change from study entry to week 48 or week 96 was calculated as (week 48 value or week 96 value) / (study entry value). Results identified above or below the limit of quantification were imputed at the quantification limit of the respective assay.
Time Frame: Study entry, weeks 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold change
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 106 | 109
Fold change
  Fold change from study entry to week 48 | 0.75 [0.44 to 1.54] | 0.88 [0.40 to 1.75] | 0.78 [0.32 to 1.54]
  Fold change from study entry to week 96 | 0.85 [0.45 to 1.64] | 0.78 [0.32 to 1.54] | 1.31 [0.65 to 2.60]

23. Secondary Outcome: Fold Change in Interleukin-6 (IL-6) From Study Entry to Weeks 48 and 96
Description: IL-6 was measured at study entry and weeks 48 and 96 (unit of measure pg/ml). Fold change from study entry to week 48 or week 96 was calculated as (week 48 value or week 96 value) / (study entry value). Results identified above or below the limit of quantification were imputed at the quantification limit of the respective assay.
Time Frame: Study entry, weeks 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold change
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 109 | 106 | 109
Fold change
  Fold change from study entry to week 48 | 0.62 [0.39 to 1.16] | 0.71 [0.51 to 1.23] | 0.75 [0.46 to 1.37]
  Fold change from study entry to week 96 | 0.89 [0.56 to 1.45] | 0.82 [0.51 to 1.34] | 0.89 [0.58 to 1.65]

24. Secondary Outcome: Fold Change in Soluble CD14 From Study Entry to Weeks 48 and 96
Description: Soluble CD14 was measured at study entry and weeks 48 and 96 (unit of measure ng/ml). Fold change from study entry to week 48 or week 96 was calculated as (week 48 value or week 96 value) / (study entry value). Results identified above or below the limit of quantification were imputed at the quantification limit of the respective assay.
Time Frame: Study entry, weeks 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold change
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 108 | 106 | 108
Fold change
  Fold change from study entry to week 48 | 1.01 [0.90 to 1.14] | 0.91 [0.78 to 1.07] | 1.00 [0.83 to 1.13]
  Fold change from study entry to week 96 | 0.98 [0.83 to 1.18] | 0.90 [0.76 to 1.02] | 0.98 [0.79 to 1.17]

25. Secondary Outcome: Fold Change in Soluble CD163 From Study Entry to Weeks 48 and 96
Description: Soluble CD163 was measured at study entry and weeks 48 and 96 (unit of measure ng/ml). Fold change from study entry to week 48 or week 96 was calculated as (week 48 value or week 96 value) / (study entry value). Results identified above or below the limit of quantification were imputed at the quantification limit of the respective assay.
Time Frame: Study entry, weeks 48 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold change
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 104 | 101 | 102
Fold change
  Fold change from study entry to week 48 | 0.54 [0.44 to 0.71] | 0.62 [0.48 to 0.78] | 0.61 [0.49 to 0.78]
  Fold change from study entry to week 96 | 0.51 [0.40 to 0.66] | 0.56 [0.43 to 0.72] | 0.58 [0.44 to 0.80]

26. Secondary Outcome: Fold Change in Percent Expression of CD38+HLADR+ on CD4+ (Percent) From Study Entry to Weeks 24 and 96
Description: Percent expression of CD38+HLADR+ on CD4+ was measured at study entry and weeks 24 and 96 (unit of measure percent). Fold change from study entry to week 24 or week 96 was calculated as (week 24 value or week 96 value) / (study entry value).
Time Frame: Study entry, weeks 24 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold change
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 101 | 95 | 101
Fold change
  Fold change from study entry to week 24 | 0.49 [0.35 to 0.70] | 0.51 [0.37 to 0.68] | 0.52 [0.40 to 0.79]
  Fold change from study entry to week 96 | 0.38 [0.24 to 0.55] | 0.34 [0.23 to 0.54] | 0.37 [0.25 to 0.56]

27. Secondary Outcome: Fold Change in Percent Expression of CD38+HLADR+ on CD8+ (Percent) From Study Entry to Weeks 24 and 96
Description: Percent expression of CD38+HLADR+ on CD8+ was measured at study entry and weeks 24 and 96 (unit of measure percent). Fold change from study entry to week 24 or week 96 was calculated as (week 24 value or week 96 value) / (study entry value).
Time Frame: Study entry, weeks 24 and 96
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Fold change
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 101 | 95 | 101
Fold change
  Fold change from study entry to week 24 | 0.51 [0.39 to 0.63] | 0.56 [0.46 to 0.71] | 0.59 [0.39 to 0.74]
  Fold change from study entry to week 96 | 0.35 [0.27 to 0.50] | 0.36 [0.24 to 0.46] | 0.38 [0.22 to 0.56]

ADVERSE EVENTS:
Description: Adverse events were not collected in this study. Please refer to the ACTG A5257 study (NCT00811954) ClinicalTrials.gov records for all adverse event summaries.
Arm/Group | Cohort A: ATV/RTV + FTC/TDF | Cohort B: RAL + FTC/TDF | Cohort C: DRV/RTV + FTC/TDF
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.